CLINICAL TRIAL: NCT02152813
Title: Efficacy of Bilateral Stimulation With Task-oriented Training in Improving Lower Limb Motor Functions in Patients With Stroke: a Randomized, Placebo-controlled Clinical Trial
Brief Title: Efficacy of Bilateral Stimulation With Task-oriented Training in Improving Lower Limb Motor Functions in Patients With Stroke
Acronym: RCT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The Hong Kong Polytechnic University (Other)
Responsible Party: Principal Investigator, Shamay Ng, Associate Professor, The Hong Kong Polytechnic University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2014_GRF_NG
Record Dates: First submitted 2014-05-29; First posted 2014-06-02 (Estimated); Last update posted 2019-03-08 (Actual); Status verified 2019-03

CONDITIONS: Stroke
Keywords: Electrical stimulation, exercise, stroke , rehabilitation
MeSH Terms: conditions — Stroke; Motor Activity | interventions — Transcutaneous Electric Nerve Stimulation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1. Bilateral TENS (Bi-TENS) group (Active Comparator): Subjects having bilateral electrical stimulation and task-orientated exercises
  Interventions: Behavioral: TENS and Task-orientated training
- Unilateral TENS (Uni-TENS) group (Placebo Comparator): Subjects having unilateral TENS over their affected lower limb only, and task-oriented exercises
  Interventions: Behavioral: TENS and Task-orientated training

INTERVENTIONS:
Behavioral: TENS and Task-orientated training — All subjects will undergo 16 sessions of their assigned intervention (60 minutes, twice a week, for 8 weeks). All subjects will receive 60 minutes task-oriented lower limb training (TOT) with electrical stimulation protocol assigned concurrently:

SUMMARY:
This proposed study aims to compare the effects of unilateral and bilateral transcutaneous electrical nerve stimulation (TENS). It will compare the effectiveness of bilateral TENS + task-oriented training (TOT) with unilateral TENS+TOTin improving muscle strength, co-ordination, dynamic standing balance, walking performance, and functional mobility in patients with chronic stroke.

The null hypothesis will be that bilateral TENS+TOT and unilateral TENS+TOT are not significantly different in promoting the recovery of these functions.

DETAILED DESCRIPTION:
This proposed study aims to compare the effects of unilateral and bilateral transcutaneous electrical nerve stimulation (TENS). It will compare the effectiveness of bilateral TENS + task-oriented training (TOT) with unilateral TENS+TOTin improving muscle strength, co-ordination, dynamic standing balance, walking performance, and functional mobility in patients with chronic stroke.

The null hypothesis will be that bilateral TENS+TOT and unilateral TENS+TOT are not significantly different in promoting the recovery of these functions.

ELIGIBILITY:
Inclusion Criteria:

* Subjects will be recruited from local self-help groups through poster advertising. \
* Subjects will be included if they (1) are between 55 and 85 years of age
* Have been diagnosed with ischaemic brain injury or intracerebral hemorrhage by MRI or computed tomography within the previous 1 to 10 years
* Are able to walk 3 metres independently with or without a walking aid
* Are able to score > 6 out of 10 on the abbreviated mental test
* Are able to follow instructions and give informed consent
* Have no skin allergy which would prevent electrical stimulation.

Exclusion Criteria:

* Subjects will be excluded if they have any additional medical, cardiovascular or orthopedic condition that would hinder proper treatment or assessment
* Use a cardiac pacemaker
* Have receptive dysphasia
* Have significant lower limb peripheral neuropathy (e.g. diabetic polyneuropathy)
* Are involved in drug studies or other clinical trials.

Ages: 55 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2014-05 (Actual); Primary Completion 2018-01 (Actual); Study Completion 2018-01 (Actual)

PRIMARY OUTCOMES:
Muscle strength of lower limb | 4 years
  The strength of maximum isometric voluntary contraction of the subject's knee extensors and flexors, ankle dorsiflexors, and plantarflexors (in kilograms) will be measured bilaterally using a Nicholas handheld dynamometer (model 01,160, Lafayette Instrument Company, Lafayette, IN) with standardized testing positions and dynamometer placement. Good to excellent reliability (ICC range, 0.84 -0.99) has been reported for lower-limb hand-held dynamometer strength measurements of subjects with neurologic conditions [49]. Each subject will complete three trials in which maximal force is generated for 2 to 3 seconds ffrom each muscle. The average of the three readings will be used for data analysis.

SECONDARY OUTCOMES:
Dynamic standing balance | 4 years
  The step test (ST) will be used to measure dynamic standing balance of both the paretic and normal limbs. It measures the number of times a subject is able to place one foot on a step 7.5cm high and back to the ground, as fast as possible, within 15 seconds. Three trials will be performed with each leg, with 1 minute of rest between trials to minimize fatigue. ST scores show excellent intra-rater and inter-rater reliability with subjects with chronic stroke.

OTHER OUTCOMES:
Lower-extremity motor coordination | 4 years
  The lower-extremity motor coordination test (LEMOCOT) will be used to measure the coordination of both the paretic and normal legs [50]. The LEMOCOT has been demonstrated as having good reliability (ICC=0.83-0.88) for subjects with subacute stroke [50]. Two red flat targets will be secured on the floor 30cm apart. The test will be performed while the subject is seated on a chair without armrests, with the knees flexed at close to 90o, the feet resting flat on the floor, and the heels on one of the targets. The subject will be instructed to touch the 2 targets alternately with the big toe, as quickly and as accurately as possible, for 20 seconds. The number of times each target is touched will be counted. The first trial will be a practice trial, with the average of the second and third trials used for analysis.

CONTACTS AND LOCATIONS:
Locations (1):
- The Hong Kong Polytechnic University, Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Kwong PWH, Ng GYF, Chung RCK, Ng SSM. Bilateral Transcutaneous Electrical Nerve Stimulation Improves Lower-Limb Motor Function in Subjects With Chronic Stroke: A Randomized Controlled Trial. J Am Heart Assoc. 2018 Feb 8;7(4):e007341. doi: 10.1161/JAHA.117.007341. PMID 29437598